CLINICAL TRIAL: NCT06086574
Title: Developing Circulating and Imaging Biomarkers Towards Personalised Radiotherapy in Lung Cancer
Acronym: VIGILANCE
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Manchester (Other)
Collaborators: Cancer Research UK (Other)
Responsible Party: Principal Investigator, CFaivreFinn, Professor Corinne Faivre-Finn, University of Manchester
Other Study IDs: NHS001986; 299279 (Other: IRAS ID); 22/NW/0297 (Other: REC number)
Record Dates: First submitted 2023-09-28; First posted 2023-10-17 (Actual); Last update posted 2023-10-17 (Actual); Status verified 2023-10

CONDITIONS: Lung Cancer Stage III
Keywords: Non small cell lung cancer; NSCLC; Stage III; Radiotherapy; Biomarker; Circulating-tumour DNA; Radiomics; PROM
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Circulating-tumour DNA is collected for analysis
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients diagnosed with stage 3 NSCLC: Patients will receive standard of care curative-intent radiotherapy treatment as decided by their primary oncologist. This includes radical radiotherapy, sequential chemoradiotherapy and concurrent chemoradiotherapy +/- consolidation immunotherapy.
  No changes in treatment. Patients will have data collected at baseline, during radiotherapy and for one year following radiotherapy. This longitudinal collection will include blood for circulating-tumour DNA analysis, electronic PROMS and radiomic analysis of standard of care imaging.

SUMMARY:
In stage 3 NSCLC, treatment and follow-up are generally performed in a 'one-size-fits-all' manner. In the setting of metastatic lung cancer there has been considerable success identifying biomarkers, which allow treatments to be tailored and lead to more personalised medicine. In patients with stage 3 disease there exists a significant unmet clinical need for equivalent biomarkers to guide treatment decisions such as to identify poor responders, predict benefit from treatment and diagnose relapse before standard of care imaging. Recent advances have made it possible to detect and quantify circulating-tumour DNA in peripheral blood of patients with stage 3 NSCLC, a promising prognostic biomarker and a measure of minimal residual disease. In addition, the information contained in routine medical images and electronic patient reported outcome measure (ePROM) questionnaires can add further predictive power to circulating tumour DNA and other clinical factors to determine patient's outcome. There is scope to integrate biomarkers in treatment decision algorithms aiming to make personalised treatment modifications (e.g. decision to treat with immunotherapy or not). VIGILANCE is a highly exploratory observational study to understand how these biomarkers might inform a future hypothesis driven interventional study.

ELIGIBILITY:
Inclusion criteria:

* Histological or cytologically confirmed NSCLC.
* Unsuitable for surgery due to tumour or patient factors.
* Stage 3 A, B or C (TNM version 8).
* Planned to receive radical radiotherapy OR sequential chemoradiotherapy OR concurrent chemoradiotherapy +/- consolidation immunotherapy.
* Predicted life expectancy >12 weeks.
* Ability to provide written informed consent.
* Willingness to comply with study procedures.

Exclusion criteria:

* Mixed non-small cell and small cell tumours.
* Adjuvant radiotherapy post-surgery.
* Participation in a study of an interventional study as part of lung cancer treatment.
* Recent/active malignant disease which might impact study results.
* Psychotic disorders/cognitive impairment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients treated under The Christie NHS Foundation Trust, Greater Manchester
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2023-03-24 (Actual); Primary Completion 2024-09-24 (Estimated); Study Completion 2025-09-24 (Estimated)

PRIMARY OUTCOMES:
Prognostic model built using baseline and longitudinal circulating-tumour DNA, radiomic features and patient reported measures to predict survival, tumour control and early tumour relapse. | 2.5 years

SECONDARY OUTCOMES:
Longitudinal description of circulating-tumour DNA patterns at baseline, during and for up to 1 year following completion of radiotherapy. | 2.5 years
Longitudinal description of radiomic features at baseline, during and for up to 1 year following completion of radiotherapy. | 2.5 years
Longitudinal description of patient reported outcomes at baseline, during and for up to 1 year following completion of radiotherapy. | 2.5 years
Predictive model built using baseline and longitudinal circulating-tumour DNA and radiomic features to predict benefit from consolidation immunotherapy. | 2.5 years
Associations between features and changes in features over time will be described, e.g. radiomic features associated with circulating-tumour DNA and radiomic features. | 2.5 years

CONTACTS AND LOCATIONS:
Locations (1):
- The Christie NHS Foundation Trust, Manchester, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided